CLINICAL TRIAL: NCT01936051
Title: Modeling Between Plasma Concentration and Serotonin Transporter Occupancy Induced by Escitalopram in Obsessive-compulsive Disorder(OCD) Patients
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jun Soo Kwon, Modeling Between Plasma Concentration and Serotonin Transporter Occupancy Induced by Escitalopram in OCD Patients, Seoul National University Hospital
Other Study IDs: H-1109-086-378; 2011-0931 (Other: Seoul National university Hospital IRB)
Record Dates: First submitted 2013-08-27; First posted 2013-09-05 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: OCD

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OCD patients: OCD patients being treated with any dose of escitalopram

SUMMARY:
To modeling the pharmacokinetic-pharmacodynamic(PK-PD) simulation with the plasma concentration and the transporter occupancy from OCD patients treated with escitalopram.

To examine the effect of G2677T/A single nucleotide polymorphism(SNP) of ABCB1 gene to the PK-PD modeling in OCD patients treated with escitalopram.

DETAILED DESCRIPTION:
To measure plasma concentration of escitalopram in OCD patients treated with escitalopram.

To measure serotonin transporter occupancy by escitalopram in OCD patients treated with escitalopram.

To genotype G2677T/A SNP of ABCB1 gene in OCD patients treated with escitalopram.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OCD based on Diagnostic and Statistical Manual(DSM)-IV criteria
* no change of escitalopram dosage in 6 weeks

Exclusion Criteria:

* psychiatric comorbidity other than OCD
* History of head injury, epilepsy, other general medical disorder

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: OCD patients
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-02; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
serotonin transporter occupancy | 72hr after oral administration of escitalopram

SECONDARY OUTCOMES:
genotype | baseline
Yale-Brown Obsessive Compulsive Scale(Y-BOCS) Score | baseline
  scale for the severity of Obsessive-compulsive symptoms
serotonin transporter occupancy | within the first 24hrs after oral administration of escitalopram
  serotonin transporter occupancy measured at 5 hour and 24 hour after oral dose of escitalopram
escitalopram plasma concentration | within 72 hours after oral administration of escitalopram
  plasma concentration of escitalopram at baseline, 1, 2, 3, 5, 8, 10, 24, 48, 72 hour after oral dose of escitalopram

CONTACTS AND LOCATIONS:
Overall Officials: Jun Soo Kwon, M.D, Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea